CLINICAL TRIAL: NCT02968719
Title: Phase 1 Pharmacokinetic (PK) Study to Evaluate Once-weekly Corplex™ Donepezil Transdermal Delivery System Compared to Daily Oral Administration of Aricept® in Healthy Adult Subjects
Brief Title: A Phase 1, Corplex™ Donepezil Transdermal System Compared to Oral Aricept®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corium, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-15086
Record Dates: First submitted 2016-11-13; First posted 2016-11-21 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (5):
- Donepezil TDS Version A (Experimental): Lead-in of 5 mg/day donepezil of target dose (1 x Corplex 5 mg donepezil transdermal delivery system; 7 days) followed by; Target dose of 10 mg/day donepezil (Treatment A); Corplex 10 mg donepezil transdermal delivery system.
  1x patch will be worn for 7 days. A total of 4 TDS patches will be applied for 4 consecutive 7 day periods.
  Interventions: Drug: Donepezil TDS Version B; Drug: Aricept
- Donepezil TDS Version B (Experimental): Lead-in of 5 mg/day donepezil of target dose (1 x Corplex 5 mg donepezil transdermal delivery system; 7 days) followed by; Target dose of 10 mg/day donepezil (Treatment B); Corplex 10 mg donepezil delivery transdermal system.
  1x patch will be worn for 7 days. A total of 4 TDS patches will be applied for 4 consecutive 7 day periods.
  Interventions: Drug: Donepezil TDS Version A; Drug: Aricept
- 10 mg Aricept (Active Comparator): 5 mg/day oral Aricept, once daily for 7 days followed by; 10 mg/day Aricept once daily for 28 days
  Interventions: Drug: Donepezil TDS Version A; Drug: Donepezil TDS Version B
- Donepezil TDS Version D (Experimental): Target dose of 5 mg/day donepezil (Treatment D) Corplex 5 mg Donepezil TDS applied for a duration of 1 week.
  Interventions: Drug: Donepezil TDS Version D; Drug: Donepezil TDS Version E
- Donepezil TDS Version E (Experimental): Target dose of 5 mg/day donepezil (Treatment E) Corplex 5 mg Donepezil TDS applied for a duration of 1 week
  Interventions: Drug: Donepezil TDS Version D; Drug: Donepezil TDS Version E

INTERVENTIONS:
Drug: Donepezil TDS Version A — Donepezil Hydrochloride Transdermal Delivery System (5mg and 10 mg Version B)
  Arms: 10 mg Aricept; Donepezil TDS Version B
Drug: Donepezil TDS Version B — Donepezil Hydrochloride Transdermal Delivery System (5 mg and 10 mg Version B)
  Arms: 10 mg Aricept; Donepezil TDS Version A
Drug: Aricept — Aricept (5 mg and 10 mg) Donepezil Hydrochloride
  Other Names: Aricept Tablet
  Arms: Donepezil TDS Version A; Donepezil TDS Version B
Drug: Donepezil TDS Version D — Donepezil Hydrochloride Transdermal Delivery System (5 mg Version D)
  Arms: Donepezil TDS Version D; Donepezil TDS Version E
Drug: Donepezil TDS Version E — Donepezil Hydrochloride Transdermal Delivery System (5 mg Version E)
  Arms: Donepezil TDS Version D; Donepezil TDS Version E

SUMMARY:
A Phase 1, Randomized, Open-Label, 3-Way Crossover, Pilot, Pharmacokinetic Study to Evaluate the Steady State Pharmacokinetics of a Once-Weekly Application of Corplex Donepezil Transdermal Delivery System (TDS) Compared to Daily Oral Administration of Aricept in Healthy Adult Subjects

DETAILED DESCRIPTION:
Part A:

60 male and female subjects will be enrolled Subjects will receive 2 versions of once-weekly Corplex Donepezil TDS and QD oral Aricept; each administered for 35 days in 3 different treatment periods.

For each treatment period; Subjects will receive a lead-in dose of approximately 5 mg donepezil/day for 7 days before commencing a dose of 10 mg donepezil/day for 28 days. Blood samples for donepezil PK and red blood cell (RBC) AChEI (as a potential pharmacodynamic [PD] marker) will be collected pre-dose through Week 8.

Adhesion and skin irritation will be monitored throughout TDS Treatments. A washout period of at least 21 days between the last study drug administration (oral administration or removal of TDS, as appropriate) in each treatment period and the first application of TDS or oral drug administration, as appropriate, in the following treatment period.

Safety will be monitored throughout the study by adverse event reporting, repeated clinical and laboratory evaluations

Part B:

Up to 47 subjects male and/or female will be enrolled This is an open-label, randomized, 2-way crossover sub-study. Eligible subjects will be randomized to 1 of 2 treatment sequences prior to the first TDS application.

Subjects will receive 2 different once-weekly Corplex Donepezil TDS treatments (Treatments D and E), each administered for 1 week, in 2 different treatment periods (Treatment Period 1 and Treatment Period 2).

In each treatment period, subjects will receive a target dose of 5 mg donepezil/day for 7 days. There will be a washout period of 35 days between removal of the first TDS in Treatment Period 1 and application of the second TDS in Treatment Period 2.

Blood samples for donepezil PK will be collected pre-dose and through to Week 6 of each treatment period.

Safety will be monitored throughout the sub-study by repeated clinical, skin irritation and laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, Caucasian, male or female ≥18 years of age at screening
* Body mass index ≥ 18.0 and ≤ 32.0 kg/m2 at screening
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or electrocardiograms (ECGs), as deemed by the Investigator.
* Have a Fitzpatrick skin type of I, II or III or have skin colorimeter scores equivalent to the allowed Fitzpatrick skin type.

Key Exclusion Criteria:

* History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds (including piperidine derivatives and other cholinesterase inhibitors)
* Has intolerance to venipuncture and/or inability to comply with the extensive blood sampling required for this study or does not have suitable veins in both arms
* Potential for occupational exposure to anticholinesterase agents.
* Female subjects with a positive pregnancy test or lactating
* Positive urine drug or alcohol results
* Estimated creatinine clearance in non-elderly subjects <80 mL/min at screening and in elderly subjects (i.e., ≥55 years of age) <60 mL/min at screening
* Hemoglobin value of less than 11.5 g/dl for females, 13.0 g/dl for males at screening and first check-in
* Any of the following drugs for 28 days prior to the first dose of study drug in Treatment Period 1 and throughout the study:

  * significant inducers of cytochrome P450 (CYP) enzymes and/or P-glycoprotein
  * anti-inflammatory drugs or cyclooxygenase 2 (COX-2) analgesic
  * beta-blockers;
  * anti-fungal medications;
  * anti-histamines;
  * cholinergics and anti-cholinergics;
  * oral corticosteroids;
  * Prolia;
  * Adjuvant analgesics
* Muscle relaxants, anti-Parkinsonian or neuroleptic medications prior to the first dose of study drug
* History or presence of excessive hairy skin on application sites as deemed by the Investigator to potentially interfere with drug absorption
* History or presence of significant skin damage, diffuse skin diseases, scars, tattoos on the application sites or other skin disturbances as deemed by the Investigator to potentially interfere with drug absorption or irritation assessments
* Use of donepezil hydrochloride or related drugs within 60 days prior to the first study drug administration
* Participation in another clinical study within 60 days prior to the first study drug administration
* Clinically significant depression symptoms or suicidal ideation or behavior as determined by the investigator:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
Steady-state PK | TDS PK sampling time-points: Predose; Day 1 (hr0); Post-dose; Day 1 (hr2,6,12); Day 2-15,22 (hr0); Day 29 (hr0,3,6,12); Day 30-35 (hr0,12) Day 36 (hr0, 2,6,12); Day 37-38,41,44,47,50,54 (hr0);
  To evaluate the steady-state PK of donepezil following once weekly Corplex Donepezil TDS application compared to once-daily (QD) oral administration of Aricept.
  Aricept PK sampling time points; Day 1 (hr0,1,2,3,4,6,8,12); Day 2,8,15,22,29 (hr0); Day 35(hr0,1,2,3,4,6,8,12); Day 36-37,40,43,46,49,53 (hr0)
PK (Part B) | TDS PK sampling time-points: Predose; Day 1 (hr0); Post-dose; Day 1 (hr2,6,12); Day 2-8 (hr0,12); Day 9,10,11,13,16,19,22,26,30,36 (hr0)
  To compare the PK of 2 once-weekly Corplex Donepezil TDS treatments (target dose 5 mg donepezil/day)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 (Part A and B) | Daily during 36-day confinement period and 7 visits over the 21 day wash-out period.
  General Safety (AE and SAE as reported by subject following guidance CTCAE v4.0)
PI assessment of local skin irritation response to TDS (Part A and B) | Part A: Daily during 36-day confinement period and 7 visits over the 21 day wash-out period. Part B:Daily during 10-day confinement period and 8 visits over the 28-35 day wash-out period.
  To evaluate the safety and tolerability (including local skin irritation) of once-weekly Corplex Donepezil TDS. Skin irritation assessed using 8 pt categorical scale based on former FDA.gov/ohrms/dockets/98fr/990236GD.pdf. The Skin Irritation scale is: no irritation; minimal erythema/barely perceptible; definite erythema readily visible, minimal edema or minimal papular response; erythema and papules; definite edema; erythema, edema and papules; vesicular eruption; strong reaction spreading beyond application site.
PI assessment of TDS Adhesion per FDA UCM504157 | Twice daily during 36-day confinement period
  To evaluate the adhesion of once-weekly Corplex Donepezil TDS. Adhesion is based on the adhered area (%) of the patch according to FDA.gov/downloads/Drugs/GuidanceComplianceRegulatory Information/Guidances/UCM504157.pdf. Specifically: ≥ 90% adhered (essentially no lift off skin); ≥ 75% to <90% adhered (some edges only lifting off skin); ≥ 50% to <75% adhered (less than half the TDS lifting off skin); < 50% adhered but did not detach (not detached, but more than half of the TDS lifting off skin without falling off); patch completely detached (TDS detached, completely off skin).

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Armas, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
No Plans